CLINICAL TRIAL: NCT03133507
Title: Effects of Reappraisal, Reassurance, and Distraction on Pain and Distress in Children Undergoing Treatment for Cancer
Brief Title: Emotion Regulation and Pain in Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Michelle Fortier, Assistant Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UCCRCC-53097
Record Dates: First submitted 2017-04-23; First posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Cancer
Keywords: cancer; salivary alpha amylase; pain; positive affect; emotion regulation strategies
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reapprasial Condition (Experimental): Children in this condition will be instructed to think about how the procedure will help them become adjusted to cold weather.
  Interventions: Behavioral: Reapprasial Condition
- Reassurance Condition (Experimental): Children will receive empathic support from the experimenter.
  Interventions: Behavioral: Reassurance Condition
- Distraction Condition (Experimental): Children in this condition will be instructed to focus their attention on a picture on a computer screen rather than on the pain.
  Interventions: Behavioral: Distraction Condition

INTERVENTIONS:
Behavioral: Reapprasial Condition — Children in this condition will be instructed to think about how the procedure will help them become adjusted to cold weather.
  Arms: Reapprasial Condition
Behavioral: Reassurance Condition — Children will be reassured by the experimenter .
  Arms: Reassurance Condition
Behavioral: Distraction Condition — Children in this condition will be instructed to focus their attention on a picture on a computer screen rather than on the pain.
  Arms: Distraction Condition

SUMMARY:
This study tested the effects of emotion regulation strategies (reappraisal, reassurance, and empathy) on pain responses in children with cancer. Children with cancer were randomly assigned to one emotion regulation strategy during an experimental pain task (the cold pressor task [CPT]). During the CPT, children rated their pain and provided saliva samples immediately before, after, and then 15 minutes after the CPT. This study examined the influence of emotion regulation on self-reported pain and physiological activity assessed through saliva samples.

DETAILED DESCRIPTION:
More than 12,000 children are diagnosed with cancer in the United States each year and the majority of these children will experience pain throughout their illness. Children with cancer are required to undergo repeated invasive medical procedures, including bone marrow aspirations (BMA) and lumbar punctures (LP), which have been described by children as the most distressing and painful aspect of their illness. The experience and memory of procedural pain can have a lasting effect and impact distress in future procedures; children learn to anticipate pain and show increased distress and decreased cooperation at subsequent procedures. Moreover, childhood medical distress has also been linked to adults' reports of pain and fear around medical events and even avoidance of future health care. Early painful procedures have also been associated with behavioral changes to medical events later in life, a finding that is supported by recent physiological evidence indicating that activation of the pain processing system in the brain can change neuropathways, which leads to increased sensitivity to later stimulation of pain systems. Therefore, it is vital to develop strategies to minimize the pain and distress that children undergo through cancer treatment and understanding the impact of children's memory on pain is a crucial step in this process.

To address this important need, this study involved identifying the strategies that children use to cope with distress that promote positive memories of medical events, examining how these strategies impact their immediate physiology (via salivary biomarkers) and self-reported pain, and understanding how these coping strategies change children's distress over time during future medical procedures. Specifically, certain coping strategies change the way that children interpret stressful medical procedures, which affects the emotional response to future procedures. These objectives were accomplished by the following specific aims:

Aim 1: Identify emotion-regulation (i.e., coping) strategies that promote more positive memories of distressing medical procedures in children with cancer.

Aim 2: Assess the impact of emotion-regulation strategies on children's distress response to painful procedures over time.

This project will provide specific means for impacting children's pain and distress during medical procedures. Specifically, because the emotion regulation strategies described in this protocol are modifiable and teachable, they provide direct implications for clinical practice in pain management by identifying strategies that can decrease children's pain and anxiety throughout their course of cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 6-18 years who were currently undergoing outpatient treatment for cancer and who could speak, read, and write in English or Spanish were eligible for the study.

Exclusion Criteria:

* Cognitive impairment, such as a developmental delay or mental retardation that would prevent children from participating in the experimental pain task.
* Children whose medical status require inpatient hospitalization or otherwise signify health complications that would prevent participation will not be recruited. Accordingly, all potential participants will be obtained via consultation with the Attending Oncology physician and/or nursing team.
* Following safety guidelines, participants will be excluded if they have a cut or sore on their non-dominant hand, have high blood pressure, or have a history of upper extremity vascular disease, cardiovascular disorder, fainting, seizures, frostbite, or chronic pain (pain lasting for more than 4 months).
* Because cortisol measures will be taken, participants will be asked to refrain from eating 1 hour before the experiment, as this can affect cortisol sample readings. In addition, because oral contraceptives can impact cortisol, participants taking hormone medications will be excluded from participation.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2012-11-14 (Actual); Primary Completion 2013-09-26 (Actual); Study Completion 2013-09-26 (Actual)

PRIMARY OUTCOMES:
Pain Tolerance | 4 mins
  Time of hand removal from the cold pressor task was recorded and used to operationally define pain tolerance with longer durations reflecting greater pain tolerance. A four-minute ceiling was used such that children were instructed to remove their hand from the water after four-minutes if they had not already done so.
Change in Salivary Alpha-Amylase | Immediately before, immediately after, and then 15 minutes after the cold pressor task.
  Salivary alpha-amylase levels (a marker of autonomic nervous system activation) was assessed using the provided saliva samples.
Self-reported pain | The exact time that participants removed their hands from water, which can range from 0-4 minutes.
  Children were asked to report their pain when they removed their hand from the water using a numeric rating scale (NRS). Children ages 6 through 11 were asked "How much is it hurting right now?" on a scale of "Not hurting" = 0 to "Hurting a whole lot" = 10. Children 12 to 18 were asked "How much pain are you in right now?" on a scale of "No Pain at All" = 0 to "A Lot of Pain" = 10.
Memory for pain | One week after the cold pressor task
  Self-reported measure of how much their hand hurt during the cold pressor task.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Fortier, Principal Investigator — 505 S. Main Street Suite 940, Orange, Ca 92868

IPD SHARING:
Plan to Share IPD: No